CLINICAL TRIAL: NCT01914263
Title: Phase 1 Study of Cord Blood-derived Cytokine-induced Killer Cells in Patients With Solid Tumor After Radical Resection
Brief Title: Safety Study of Cord Blood-derived Cytokine-induced Killer Cells in Patients With Solid Tumor After Radical Resection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alliancells-PuRui Biocience Co., Ltd. (Industry)
Collaborators: Zhongyuan Union Stem Cell Bio-engineering Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlliancellsPuRui-01
Record Dates: First submitted 2013-07-29; First posted 2013-08-02 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2014-07

CONDITIONS: Hepatocellular Carcinoma; Renal Cell Carcinoma; Lung Cancer
Keywords: Cord blood-Derived cytokine induced killer cells,; Radical resection
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cytokine induced killer cell (Experimental): The eligible patients are infused a single dose of 8x10^9 CIK cells.
  Interventions: Biological: cytokine induced killer cell
- Control (No Intervention): The eligible patients are followed up for 30 days without any treatment.

INTERVENTIONS:
Biological: cytokine induced killer cell — The eligible patients are infused with a single dose of 8x10^9 cord blood-derived cytokine indued killer cells.
  Arms: cytokine induced killer cell

SUMMARY:
Cytokine-induced killer (CIK) cells are a heterogeneous subset of ex-vivo expanded T lymphocytes which present a mixed T-NK phenotype and are endowed with a major histocompatibility complex-unrestricted antitumor activity. Radical surgery is a good therapy for patients with solid tumor.However, tumor relapse is still a risk for those patients. Our hypothsis is that cytokine induced killer cells maybe decrease the recurrence rate. The purpose of this study is to evaluate the safety and tolerability of cord blood-derived cytokine induced killer cells in patients with solid tumor following radical resection.

DETAILED DESCRIPTION:
It was estimated that 2.6 million people suffer from cancer and 1.8 million die of cancer in China yearly according to the Annual Report of Cancer Registration in China 2012. So far, the main treatment modalities for tumors have been surgery, radiotherapy and chemotherapy. However, tumor relapse is still a risk for those patients underwent the conventional therapy. With the development of oncology and immunology in recent years, immunotherapy represents a novel path to obtain a durable and long-lasting response in cancer patients. Cytokine-induced killer (CIK) cells are a heterogeneous subset of ex-vivo expanded T lymphocytes which present a mixed T-NK phenotype and are endowed with a MHC-unrestricted antitumor activity. CIK cells are expanded conventionally from peripheral blood mononuclear cells by addition of a variety of cytokines in vitro culture.

Autologous CIK cells infusion therapy for patients with malignancies is reported world widely. However, there are several drawbacks for autologous CIK limiting its clinical application. For example, limited cell numbers, decreased cell activities, and unavailable in time etc. Cord blood, as a novel source of non-senescent lymphocytes for tumor immunotherapy, has been focused on recently. Accumulating preclinical studies have shown that cord blood-derived CIK cells are potent anti-tumor effectors using in adoptive cancer immunotherapy. However it is unclear whether administration of cord blood-derived CIK cells is safe in patients with malignancies. Our previous studies demonstrated that clinical scale expansion of CIK from cord blood is feasible. The cord blood-derived CIK cells exhibit antitumor effect in vitro and in vivo (tumor bearing nude mice) against a variety of tumor cells including ZR751, MCF7, HepG2, SMMC-7721, Hela, A375, DU145, H1299 and A549. Furthermore, intravenous infusion of a single dose of 3X10^8 cord blood-derived CIK cells in mice is safe.

The purpose of this study is to evaluate the safety and tolerability of cord blood-derived CIK cells in patients with solid tumor following radical resection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over 18 years of age.
* Patients who give written informed consent.
* Patients with solid tumor already had radical resection
* Definition of radical resection in this study:
* All tumors were moved out, with a clean resection margin.
* No distance metastasis.
* No major post-operative complication.
* Without any anti-cancer medication within the past 15 days.
* The following laboratory parameters: Platelet count >= 70 x 109/L; Hemoglobin >= 8.5 g/dL; Albumin >= 3.5 g/dL; Total bilirubin <= 25umol/L; Alanine transaminase (ALT) and AST <= 2.5 x upper limit of normal; Serum creatinine <= 1.5 x the upper limit of normal; Prothrombin time (PT) <= 3 seconds above control.

Exclusion Criteria:

* History of cardiac disease.
* Active clinically serious infections
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* History of organ allograft.
* Known or suspected allergy to the investigational agent or any agent given in association with this trial.
* Pregnant or breast-feeding patients.
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study.
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events following infusion of cord blood-derived cytokine-induced killer cells. | 30 days post-infusion
  The primary outcome measures for safety will include the incidence of fever,chill,rash and Graft-versus-Host Disease (GVHD).

SECONDARY OUTCOMES:
Haematology | Baseline, 1 day, 3 days 10 days and 30 days after cell infusion
  These parameters include erythrocytes, leukocytes, platelets, T cell, B cell, Natural killer cell, CD4/CD8, Th1/Th2, Th17 cell and Treg cell.
Serological analysis | Baseline, 1day, 3 days 10 days and 30 days after cell infusion
  immunoglobulin G, immunoglobulin A, immunoglobulin D, immunoglobulin E and immunoglobulin M. Albumin (ALB), Alanine aminotransferase (ALT), Aspartate Aminotransferase (AST), Prealbumin(PA), total bilirubin (TB), and direct bilirubin (DB); Blood urea nitrogen(BUN), Urea (UA), and Crea (Cr); Total cholesterol (TC), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C), triglycerides (TG), very low density lipoprotein cholesterol (VLDL-C), and Non-HDL-C; blood sugar;

CONTACTS AND LOCATIONS:
Overall Officials: mingyuan wu, MD, Study Chair
Locations (3):
- China (3):
  - Hannan BOAO Life infinity international anti-aging medical center, Qionghai, Hainan
  - The 210 Hospital of Chinese People's Liberation Army, Dalian, Liaoning
  - The 323 Hospital of Chinese People's Liberation Army, Xi'an, Shaanxi